CLINICAL TRIAL: NCT00000967
Title: Safety and Tolerance of Zidovudine and Interferon-Alpha in HIV-Infected Children
Brief Title: The Safety of Zidovudine Plus Interferon-Alpha in HIV-Infected Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Glaxo Wellcome (Industry); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 153; 11128 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; AIDS-Related Complex; Zidovudine; Interferon Type I
MeSH Terms: conditions — HIV Infections; AIDS-Related Complex | interventions — Interferon alpha-2; Zidovudine

INTERVENTIONS:
Drug: Interferon alfa-2a
Drug: Zidovudine

SUMMARY:
PRIMARY: To determine the maximum tolerated dose of interferon-alfa (IFN-A) alone and in combination with zidovudine (AZT); to assess the safety and tolerance of IFN-A alone and in combination with AZT.

SECONDARY: To evaluate the effect of combination IFN-A and AZT on immunologic and virologic parameters; to determine whether the pharmacokinetic parameters of AZT are modified by the subcutaneous administration of IFN-A.

AZT is effective in suppressing the progression of HIV infection in patients without symptoms or with AIDS or AIDS-related complex (ARC). However, use of AZT is limited by its frequent toxicity, which sometimes relates to the amount of drug given. Thus, a combination treatment of two drugs that work together may provide more effective and safer treatment. IFN-A is a drug that has antiviral effects and may work well with AZT.

DETAILED DESCRIPTION:
AZT is effective in suppressing the progression of HIV infection in patients without symptoms or with AIDS or AIDS-related complex (ARC). However, use of AZT is limited by its frequent toxicity, which sometimes relates to the amount of drug given. Thus, a combination treatment of two drugs that work together may provide more effective and safer treatment. IFN-A is a drug that has antiviral effects and may work well with AZT.

The study is being conducted in three stages. In Cohort A (IFN-A alone), four patients receive IFN-A; subsequent four-patient cohorts receive doses escalated in increments. If 50 percent or more of patients at any dose level experience grade 2 or better toxicity, doses in subsequent cohorts are escalated. If grade 3 or 4 toxicity is seen in one patient at a given dose level, two additional patients are enrolled at that level. Treatment is given subcutaneously (under the skin, with a needle), 3 times per week for 12 weeks. The MTD is defined as the dose level immediately below that at which 50 percent or more of patients experience grade 3 or 4 toxicity. In Cohort B (combination IFN-A plus AZT), patients who complete treatment in Cohort A continue on the same dose of IFN-A, and a low, middle, or high dose of AZT is added. In Cohort C, four newly assigned patients who have been on a stable prescribed dose of AZT of at least 90 mg/m2 for 6 weeks are treated at each of the same dose combinations as those in Cohort B. Treatment is given for 12 weeks. IFN-A is given subcutaneously 3 times a week and AZT is given orally every 6 hours. Dose levels of both drugs are increased until 50 percent or more of patients experience grade 3 or 4 toxicity in any dose level.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Recommended:

* Prophylaxis for Pneumocystis carinii pneumonia.

Allowed:

* Aerosol ribavirin for short-term treatment of acute respiratory syncytial virus (RSV).
* Immunization according to the current recommendations of the Advisory Committee for Immunization Practice.
* IVIG. Systemic ketoconazole, acyclovir, or oral nystatin for acute therapy.

Patients must have the following:

* HIV infection. Patients with proven resistance to AZT are also eligible.

Prior Medication:

Allowed:

* Aerosol ribavirin.

Required:

Cohort C treatment:

* Stable prescribed dose of zidovudine (AZT) >= 90 mg/m2 for at least 6 weeks prior to study entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded: AIDS or class P-2B, D, or E symptomatic infection.

Concurrent Medication:

Excluded:

* Hepatotoxic or neurotoxic drugs, immunosuppressants, or antiseizure medication. Ketoconazole, fluconazole, and acyclovir for prophylaxis. Immunomodulators (other than IVIG). Experimental drugs.

Cohort A patients:

* AZT for clinical indications.

Prior Medication:

Excluded:

* Other antiretroviral agents (including didanosine (ddI), dideoxycytidine (ddC), or soluble CD4) within 1 month of study entry. Systemic ribavirin administered for retroviral therapy within 2 months of study entry.
* Immunomodulating agents including interferon, isoprinosine, interleukin-2, or lymphocyte transfusions within 4 weeks of study entry.
* RBC transfusion within 4 weeks prior to study entry.

Alcohol or drug abuse.

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52
Dates: Study Completion 1996-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diaz C, Study Chair; Yogev R, Study Chair
Locations (9):
- United States (6):
  - Cook County Hosp., Chicago, Illinois
  - Chicago Children's CRS, Chicago, Illinois
  - Tulane/LSU Maternal/Child CRS, New Orleans, Louisiana
  - BMC, Div. of Ped Infectious Diseases, Boston, Massachusetts
  - NYU Med. Ctr., Dept. of Medicine, New York, New York
  - St. Jude/UTHSC CRS, Memphis, Tennessee
- Puerto Rico (3):
  - Univ. Hosp. Ramón Ruiz Arnau, Dept. of Peds., Bayamón
  - San Juan City Hosp. PR NICHD CRS, San Juan
  - Univ. of Puerto Rico Ped. HIV/AIDS Research Program CRS, San Juan

REFERENCES:
- [Background] Diaz C, Yogev R, Culnane M, Rogers A, Van Dyke R, Fenton T. ACTG 153: a multicenter phase I study of alpha-interferon in HIV infected children. AIDS Clinical Trials Group. Int Conf AIDS. 1994 Aug 7-12;10(1):79 (abstract no 269B)
- [Background] Clemente D, Yogev R, Culnane M, Rogers A, Van Dyke R, Hetherington S, Fenton T. ACTG 153: phase I, open-label; dose escalating study of interferon-alpha alone and in combination with zidovudine in children with early HIV disease. Program Abstr Intersci Conf Antimicrob Agents Chemother. 1994 Oct 4-7:35